CLINICAL TRIAL: NCT04505696
Title: Effect of Providing Speech Therapy Awareness in Private Schools
Brief Title: Providing Speech Therapy Awareness in Private Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REC/00735 Saania Amjad
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Speech and Language Disorder; Speech Therapy; Speech Delay; Swallowing Disorder; Acquired Language Disorders; Developmental Delay Disorder; Stuttering; Hearing Impairment; Head and Neck Cancer
Keywords: Speech-Language Pathology; Awareness; Intervention; Teacher training
MeSH Terms: conditions — Speech; Language Disorders; Communication Disorders; Language Development Disorders; Deglutition Disorders; Developmental Disabilities; Stuttering; Hearing Loss; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Single group pre-post
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Speech-Language Pathology Introduction and scope (Other): Demographic Information Section on Knowledge & Awareness Section on Practices
  Interventions: Other: Speech-Language Pathology Presentation

INTERVENTIONS:
Other: Speech-Language Pathology Presentation — 45 minutes presentation on Speech-Language Pathology introduction and scope Introduction to speech and language Introduction to a range of disorders The scope of practice

SUMMARY:
There has been limited research in the area of speech and language therapy awareness in Pakistan. The study aims to assess the efficacy of providing speech therapy awareness in private schools through a pre-post model. This Quasi experimental study will be a means of reaching out to schools and directly create awareness regarding the field and its scope. Pre-assessment will be carried out and after which a 45 minutes presentation will be conducted face to face or through a webinar as per school directives. The results will be analysed quantitatively and pre-post assessment of the participants will be measured.

DETAILED DESCRIPTION:
There has been limited research in the area of speech and language therapy awareness in Pakistan. The study aims to assess the efficacy of providing speech therapy awareness in private schools through a pre-post model. the study design is Quasi Experimental study

Sample size: 385. Raosoft Sampling technique: Purposive Sampling Inclusion criteria: Private English medium schools of Islamabad and Rawalpindi. Schools with no speech and language therapists Exclusion criteria: Public Schools and schools who may have visiting or permanent speech therapists on their panel.

Delphi technique will be used for development of a tool for the intervention and to assess the impact of the awareness program.

The teachers will be tested pre and post program and three months after the completion of the program. Three months post they will be a) tested on the same questionnaire b) will determine number of students identified with difficulties c) students referred to a therapist.

Data will be analyzed quantitative means and quantitative data will be analyzed using SPSS

ELIGIBILITY:
Inclusion Criteria:

* Private English medium schools of Islamabad and Rawalpindi. Schools with no speech and language therapists

Exclusion Criteria:

* Public Schools and schools who may have visiting or permanent speech therapists on their panel

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Pre-post Questionnaire | Same 1 Day
  A reliable and valid tool will be used for assessment of Knowledge, awareness and practice regarding the speech-language pathology profession and the scope of practice. The tool consists of demographic information, comprising of 45 questions, placed under 3 sections.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha K Butt, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glover A, McCormack J, Smith-Tamaray M. Collaboration between teachers and speech and language therapists: Services for primary school children with speech, language and communication needs. Child Lang Teach Ther [Internet]. 2015 Oct 7 [cited 2020 Apr 26];31(3):363-82. Available from: http://journals.sagepub.com/doi/10.1177/0265659015603779
- [Background] Mcleod S, Mckinnon DH. Title: Support required for primary and secondary students with communication disorders and/or other learning needs Journal: Child Language Teaching and Therapy. journals.sagepub.com. 2010 Jun;26(2):123-43.
- [Background] Abdalla F, St Louis KO. Modifying attitudes of Arab school teachers toward stuttering. Lang Speech Hear Serv Sch. 2014 Jan;45(1):14-25. doi: 10.1044/2013_LSHSS-13-0012. PMID 24687764
- [Background] Kataoka M, Van Kraayenoord CE, Elkins J. Principals' and teachers' perceptions of learning disabilities: A study from Nara Prefecture, Japan. Vol. 27, Learning Disability Quarterly. SAGE Publications Inc.; 2004. p. 161-75.
- [Background] Zamani P, Hozeily E, Tahmasebi N, Ahmadi A, Moradi N. The effect of elementary school teachers' knowledge of learning disabilities on referring afflicted students to speech therapy. Iran Rehabil J. 2018 Dec 10;16(4):371-7.
- [Background] Kakabaraee K, Arjmandnia A, and GA-P-S, 2012 undefined. The study of awareness and capability of primary school teachers in identifying students with learning disability in the province of Kermanshah. Elsevier [Internet]. [cited 2020 May 3]; Available from: https://www.sciencedirect.com/science/article/pii/S1877042812016631
- [Background] McNeill BC, Gillon GT, Dodd B. Effectiveness of an integrated phonological awareness approach for children with childhood apraxia of speech (CAS). Child Lang Teach Ther [Internet]. 2009 Oct 26 [cited 2020 Apr 26];25(3):341-66. Available from: http://journals.sagepub.com/doi/10.1177/0265659009339823
- [Background] Abrahams K, Harty M, St Louis KO, Thabane L, Kathard H. Primary school teachers' opinions and attitudes towards stuttering in two South African urban education districts. S Afr J Commun Disord. 2016 Jul 27;63(1):e1-e10. doi: 10.4102/sajcd.v63i1.157. PMID 27796099
- [Background] Mahmoud HN, Alkhamra R. A Study of Public Awareness of Speech-Language Pathology in Amman A Study of Public Awareness of Speech - Language Pathology in Amman. 2015;(December).
- [Background] Regina LB. SPEECH LANGUAGE PATHOLOGY A REWARDING PROFESSION FILLED WITH SHORTAGES. Southeast Educ Netw [Internet]. 2018 Jul 1 [cited 2020 May 2];1. Available from: https://www.seenmagazine.us/Articles/Article-Detail/ArticleId/6691/SPEECH-LANGUAGE-PATHOLOGY
- [Background] Mulcair G, Pietranton AA, Williams C. The International Communication Project: Raising global awareness of communication as a human right. Int J Speech Lang Pathol. 2018 Feb;20(1):34-38. doi: 10.1080/17549507.2018.1422023. Epub 2018 Jan 22. PMID 29355390